CLINICAL TRIAL: NCT02738918
Title: Belatacept (Nulojix) in Renal Transplant Recipient With Mild Immunologic Risk Factor: a Pilot Prospective Study
Acronym: BELACOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P121203
Record Dates: First submitted 2016-01-05; First posted 2016-04-14 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2017-11

CONDITIONS: Renal Transplant; Acute Antibody Mediated Rejection; Mild Immunologic Risk Factor
Keywords: Renal Transplant; Anti HLA antibodies; Humoral rejection
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nulojix (Experimental)
  Interventions: Drug: Nulojix (Belatacept)

INTERVENTIONS:
Drug: Nulojix (Belatacept) — Nulojix Administration will start the day of transplantation (day 1 and first dosing day);10 mg/kg : (day1, 5,14,28 ), Week 8 and 12 and then 5 mg/kg every 4 weeks until Month 12

SUMMARY:
BACKGROUND: Antibody-mediated humoral rejection is currently a critical question in renal transplant recipient with immunological risk factors such as pre transplant donor-specific anti HLA antibodies (DSA). The immunosuppressive management of the patients is still not well defined and improving both short and long-term graft outcome remains a challenging question. Recent experimental data suggest that Belatacept could induce B cell anergy , induce regulatory B cell and decrease Ig production. These findings are strengthened by the results of both phase II and III clinical studies, showing a significant lower incidence of DSA in patients treated with Belatacept compared to recipients receiving a conventional immunosuppressive regimen with calcineurin inhibitors (CNI).

Primary objective will be the incidence of clinical and subclinical humoral rejection (According to BANFF 2011 Criteria). Secondary objectives will include one-year graft and patient survival, renal function at M12 (MDRD), incidence of cellular rejection (M 12), level of proteinuria (M3 and M12) and DSA outcome (outcome of DSA MFI at JO, M3 and M12). Inclusion period will be of two years. DSA identification and quantitative analysis before and after transplantation will be centralized in only one HLA laboratory Unit (Hospital Saint Louis) for providing results homogeneity.

According to previous clinical studies, the incidence of Acute Antibody Mediated Humoral Rejection is close to 20% in patients with mild immunological risk defined by the presence of DSA at the time of transplant with mean fluorescence intensity (MFI) between 1000 and 3000 (Luminex). In order to demonstrate a significant reduction (40%) of AAMR and sAAMR incidence, 91 patients will be included in this study. Results will be compared to a cohort matched for age, sex, immunological risk factor (DSA), time of transplant, transplant center and grafted with a similar immunosuppressive regimen including CNI instead of Belatacept

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   a) Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
2. Target Population

   a) Renal transplant recipients aged over 18 with DSA at the time of transplant and or on historic serum with mean fluorescence intensity (MFI) between 500 and 3000 (Luminex), available at the time of the transplant.
3. Age and Sex

   1. Men and women, ages >18
   2. Women of childbearing potential (WOCBP) must be using two adequate methods of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of study drug to minimize the risk of pregnancy.

   WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:
   * Amenorrhea that has lasted for 12 consecutive months or more without another cause, or
   * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.

   Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

   WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of the investigational product.

   A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 8 weeks after the last dose of study drug to minimize the risk of pregnancy.

   Exclusion Criteria:
4. Sex and Reproductive Status

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of study drug.
   2. Women who are pregnant or breastfeeding.
   3. Women with a positive pregnancy test.
   4. Sexually active fertile men not using effective birth control if their partners are WOCBP.
5. Target Disease Exceptions

   1. Subjects who are EBV-negative or whose EBV status is unknown..
   2. Renal Transplantation of Focal and Segmental Glomerulosclerosis
6. Medical history and concomitant diseases
7. Patient with past history of malignancy
8. Physical and Laboratory Test Findings: DSA <500 or>3000
9. Allergies and Adverse Drug Reactions to Nulojix
10. Other Exclusion Criteria

    1. Prisoners, or subjects who are involuntarily incarcerated.
    2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Antibody Mediated Rejection (AAMR) (According to BANFF 2011 Criteria) | 12 months (+/- 3 months)

SECONDARY OUTCOMES:
Incidence of subclinical AAMR diagnosed on protocol biopsy | 3 months (+/- 1 month), 12 months (+/- 3 month)
Number of patient survival | 12 months (+/- 3 months)
Number of graft survival | 12 months (+/- 3 months)
Renal function measure by creatinine clearance (ml/min) (MDRD formula) | 3 months (+/- 1 month), 12 months (+/- 3 months)
Incidence of clinical and subclinical cellular rejection | 12 months (+/- 3 months)
Renal function by level of proteinuria (in g/l) | 3 months (+/- 1 month), 12 months (+/- 3 months)
Donor Specific Antibody (DSA) level, evaluate by the measure of maximal Mean Fluorescence Intensity (MFI)by Luminex Single Antigen | 3 months (+/- 1 month), 12 months (+/- 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRIMBERT, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Lefaucheur C, Loupy A, Hill GS, Andrade J, Nochy D, Antoine C, Gautreau C, Charron D, Glotz D, Suberbielle-Boissel C. Preexisting donor-specific HLA antibodies predict outcome in kidney transplantation. J Am Soc Nephrol. 2010 Aug;21(8):1398-406. doi: 10.1681/ASN.2009101065. Epub 2010 Jul 15. PMID 20634297
- [Background] Gaston RS, Cecka JM, Kasiske BL, Fieberg AM, Leduc R, Cosio FC, Gourishankar S, Grande J, Halloran P, Hunsicker L, Mannon R, Rush D, Matas AJ. Evidence for antibody-mediated injury as a major determinant of late kidney allograft failure. Transplantation. 2010 Jul 15;90(1):68-74. doi: 10.1097/TP.0b013e3181e065de. PMID 20463643
- [Background] Loupy A, Suberbielle-Boissel C, Hill GS, Lefaucheur C, Anglicheau D, Zuber J, Martinez F, Thervet E, Mejean A, Charron D, Duong van Huyen JP, Bruneval P, Legendre C, Nochy D. Outcome of subclinical antibody-mediated rejection in kidney transplant recipients with preformed donor-specific antibodies. Am J Transplant. 2009 Nov;9(11):2561-70. doi: 10.1111/j.1600-6143.2009.02813.x. Epub 2009 Sep 22. PMID 19775320
- [Background] Haas M, Montgomery RA, Segev DL, Rahman MH, Racusen LC, Bagnasco SM, Simpkins CE, Warren DS, Lepley D, Zachary AA, Kraus ES. Subclinical acute antibody-mediated rejection in positive crossmatch renal allografts. Am J Transplant. 2007 Mar;7(3):576-85. doi: 10.1111/j.1600-6143.2006.01657.x. Epub 2007 Jan 4. PMID 17229067